CLINICAL TRIAL: NCT07278765
Title: Optimizing Engagement With Digital Mental Health Services Among Sexual And Gender Minority Consumers
Brief Title: QT-Digital Mental Health Engagement Study
Acronym: QT-DIMES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Mental Health America (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Meghan Romanelli, Assistant Professor: School of Social Work, University of Washington
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Health Services Research
Other Study IDs: STUDY00017726; K01MH131795-01A1 (NIH)
Record Dates: First submitted 2025-12-05; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Engagement, Patient
Keywords: Digital Mental Health
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HAPA Engagement Strategies (Experimental): At each decision point in the MHA Screening Program flow, each eligible participant will be randomized to either receive a HAPA-based engagement strategy or not. Participants will be randomized with equal probability (0.2) to either receive: 1) no engagement strategy (i.e., the standard Next Steps resource page as usual; control), or; 2) one of four types of HAPA-based engagement strategies. Participants randomized to receive an engagement strategy will be randomized with equal probability to an engagement strategy targeting a HAPA construct: 1) outcome expectancy; 2) self-efficacy; 3) perceived risk, and; 4) barriers and resources. The first decision point will be the screening Results page which is displayed immediately after completing the PHQ-9 and optional demographic questions. The second decision point will be the targeted Next Steps resource page that participants click on from the Results page.
  Interventions: Behavioral: HAPA Engagement Strategies
- Results Page Comparator (No Intervention): Users see the usual MHA Results Page without engagement strategies.
- Resource Page Comparator (No Intervention): Users see the usual MHA Next Steps resource pages without engagement strategies.

INTERVENTIONS:
Behavioral: HAPA Engagement Strategies — Participants will be delivered HAPA-based engagement strategies directly on the MHA website, including on the Results page and targeted Next Steps resource page. The engagement strategies target HAPA behavioral determinants: outcome expectancy, self-efficacy, perceived risk, and barriers and resources. On the Results page, these engagement strategies will be displayed as inline messages designed to quickly reinforce a HAPA behavioral determinant before users choose their Next Steps. On the Next Steps resource page, these HAPA-based engagement strategies will be displayed as inline cards embedded directly within the page layout.
  Arms: HAPA Engagement Strategies

SUMMARY:
Sexual and gender minority (SGM) populations are disproportionately impacted by mental health concerns relative to their heterosexual and cisgender peers. Despite high need, SGM populations continue to report unmet mental health needs because they cannot or do not access mental health services. Digital Mental Health (DMH) services have been recognized as feasible, economical, and effective options to broaden the availability of mental health care to consumers who face barriers to mental health help-seeking. SGM consumers cite a preference for DMH care and this delivery format holds promise to attend to major mental health care access barriers experienced by this consumer group. Yet, the availability of DMH services tailored to the needs of SGM consumers is limited, and a dearth of research examines SGM populations' actual engagement with DMH services. A potential solution to fully understand how SGM populations utilize DMH services would be to characterize their engagement within a natural setting. Leveraging an established partnership with Mental Health America (MHA), a non-profit mental health advocacy group offering free, evidence-based screenings and self-guided DMH resources, this study will follow a large, naturalistic sample of SGM DMH consumers with the aim to test tailored engagement strategies with SGM DMH consumers using a micro-randomized trial (MRT) design. Results of this study will inform if delivering engagement strategies can meaningfully increase initial and sustained engagement with MHA resources and which types of strategies, specifically, work best for which users.

DETAILED DESCRIPTION:
This study aims to evaluate the feasibility of testing tailored engagement strategies with SGM DMH consumers using a micro-randomized trial (MRT) design and to create preliminary evidence about which theory-driven strategies most effectively promote engagement with DMH resources. This study will involve delivering brief, theory driven engagement strategies at two key decision points within the flow of MHA's Screening Program and assess feasibility of integrating these strategies into MHA's existing web infrastructure and testing them in a naturalistic setting.

The primary objective is to evaluate whether delivering (vs. not delivering) engagement strategies after an online depression screening increases initial and sustained engagement with DMH resources on the MHA website, and to understand which engagement strategy might be most effective. The engagement strategies are grounded in the Health Action Process Approach (HAPA), including immediate behavioral determinants: outcome expectancy, self-efficacy, perceived risk, and barriers and resources.

Eligibility assessment will begin after a user completes the online depression screening (PHQ-9) hosted on the MHA website as part of their Screening Program. Users who complete the online PHQ-9 and optional demographic questions will be considered for inclusion. Those who are aged 14+ and SGM will be randomized at each decision point to either receive or not receive engagement strategies. Participants will encounter two randomization decision points embedded within the usual user flow of the MHA Screening Program.

The first decision point will be the Results page where users are typically shown information about their PHQ-9 score and provided a set of 3-4 targeted Next Steps resources. Here, participants will be randomized with equal probability (0.2) to either receive: 1) no engagement strategy (i.e., the standard Results page as usual; control), or; 2) one of four types of HAPA-based engagement strategies. Participants randomized to receive an engagement strategy will be randomized with equal probability to an engagement strategy targeting a HAPA construct: 1) outcome expectancy; 2) self-efficacy; 3) perceived risk, and; 4) barriers and resources. On the Results page, these engagement strategies will be displayed as inline messages designed to quickly reinforce a HAPA behavioral determinant before users choose their Next Steps. The second decision point will be the targeted Next Steps resource page that participants click on from the Results page. Here, participants will be randomized with equal probability (0.2) to either receive: 1) no engagement strategy (i.e., the standard Next Steps resource page as usual; control), or; 2) one of four types of HAPA-based engagement strategies. Participants randomized to receive an engagement strategy will be randomized with equal probability to an engagement strategy targeting a HAPA construct: 1) outcome expectancy; 2) self-efficacy; 3) perceived risk, and; 4) barriers and resources. On the Next Steps resource page, these HAPA-based engagement strategies will be displayed as inline cards embedded directly within the page layout. These cards function as small UI components (e.g., badges) that visually stand out but do not interrupt user navigation. Each card is delivered seamlessly near the top of the Next Steps resource page content and can be read without being redirected or leaving the page.

Randomizations are independent across decision points. Delivery of engagement strategies occurs passively within the website UI and does not alter the standard navigation flow.

The primary engagement outcome will include participants' click-through to the targeted Next Steps resource and total time on the targeted Next Steps resource. Secondary engagement outcomes will include the total time on MHA pages and total number of MHA pages visited beyond the Results and targeted Next Steps resource, capped at 30 minutes of inactivity. All engagement outcomes will be captured automatically through MHA's analytics system.

ELIGIBILITY:
Inclusion Criteria:

* Users of the Mental Health America (MHA) website engaging from Internet Protocol (IP) addresses in the United States
* Completed the PHQ-9 depression screener in English
* Answered MHA's standard demographic questions that identify users as age 14 and older
* Answered MHA's standard demographic questions that identify users as LGBTQ+.

Exclusion Criteria:

* IP addresses outside of the United States
* Do not answer MHA's standard demographic questions
* Answered MHA's standard demographic questions that identify users as age 13 and younger
* Answered MHA's standard demographic questions that identify users as not LGBTQ+.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Proximal engagement | 30 minutes
  Initial engagement, i.e., click-through to the targeted Next Steps resource, capped at 30 minutes of inactivity.
Proximal engagement | 30 minutes
  Sustained engagement, i.e., total time on the targeted Next Steps resource, capped at 30 minutes of inactivity.

SECONDARY OUTCOMES:
Proximal engagement | 30 minutes
  Total time on MHA pages beyond the Results and targeted Next Steps resource, capped at 30 minutes of inactivity.
Proximal engagement | 30 minutes
  Total number of MHA pages visited beyond the Results and targeted Next Steps resource, capped at 30 minutes of inactivity.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Romanelli, PhD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Mental Health America, Alexandria, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided